CLINICAL TRIAL: NCT03190382
Title: SHOW-ME PAD (Peripheral Artery Disease)
Brief Title: SHOWME-PAD (Peripheral Artery Disease)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-053
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Received Decision Tool (Experimental): Peripheral artery disease patients that received the decision support tool.
  Interventions: Other: Decision Support Tool

INTERVENTIONS:
Other: Decision Support Tool — Patients enrolled in the study will receive the decision tool prior to the first PAD clinic visit and the medical decision making conversation with the provider.

SUMMARY:
The overall goal of SHOWME-PAD is to make the existing evidence-base on treatment outcomes -focusing on health status outcomes that reflect the patients' perspective - more transparently available to patients and providers, such that more informed, evidence-based shared treatment decisions occur. INTEGRITY-PAD has the potential to radically reorganize care delivery to patients with PAD such that more value for the patient and society will be created.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a burdensome condition that affects 10% of the population and increases to 15-20% among those ≥70 years. In PAD, the underlying pathophysiologic process, atherosclerosis, presents itself as blockages in patients' leg arteries that prevent adequate blood flow and can result in burning calf (or buttock) pain while walking and that is relieved upon rest ('intermittent claudication'). In extreme cases, PAD can progress to critical limb ischemia, characterized by ulceration, gangrene, and threatened limb viability. Patients with PAD have significant atherosclerotic risk factors and impaired health status - thus creating 2 therapeutic goals, prevention of cardiovascular events and improved symptom control and quality of life. While the onset of PAD tends not to be as abrupt as for other cardiovascular conditions, such as stroke or myocardial infarction, leg symptoms can severely affect patients' health status (their symptoms, functional status, and quality of life). In addition, patients' risk of having a cardiovascular event is disproportionately high, as compared with other cardiovascular diseases. One-year cardiovascular event rates - including cardiovascular death, myocardial infarction, or stroke, or other hospitalizations for atherothrombotic events - are estimated to be over 21% in patients with PAD, as compared with 15% for coronary artery disease and stroke.9 Mortality rates are 15-30% 5 years after diagnosis. Part of these disproportionate event rates may be explained by under recognition and under treatment of PAD and its underlying atherosclerotic process. Finally, PAD not only impacts patients' individual lives and their families; it also has a tremendous impact on society at large. It is estimated that annual costs associated with vascular-related hospitalizations in PAD patients in the US exceeds $21 billion.

The primary treatment goals for PAD are symptom relief, quality of life improvement, and cardiovascular risk reduction. Several treatment options are available for PAD, ranging from invasive revascularization procedures, including peripheral percutaneous intervention (PPI) and surgical revascularization to non-invasive options, including supervised and home-based exercise therapy, PAD-specific medications, and cardiovascular risk management. While there is no "gold-standard" treatment for PAD, less invasive options are recommended as a first-choice treatment. Despite these recommendations, invasive procedures are often first offered to patients, with no alternative options being discussed. In treatment scenarios with a lot of clinical equipoise (i.e. uncertainty about what treatment would be best) and a rapidly growing market for newly-introduced technologies, including medical devices for invasive PAD procedures (e.g. stents for endovascular treatment), with limited performance measurement and accountability criteria, there is a high risk of unwanted variation in treatment practices, misallocation of treatments, and unnecessary costs.

Given this context, some of the current challenges in current PAD care include: 1) limited access to the evidence-base in routine clinical care for patients and providers; 2) the potential mismatch of PAD treatments to patient preferences and profiles; and 3) patients not being informed or engaged in medical decision making. These challenges may leave patients uninformed about treatment risks and benefits, increase the risk of misallocating treatments to patients, and may unnecessarily increase costs. A very promising strategy to overcome these challenges is the use of evidence-based, decision support tools. Importantly, it is currently unknown whether patient-centered PAD decision-tools can be designed to improve the alignment of patients' values with respect to their treatment choice and whether these tools can improve patients' knowledge and access to the evidence-base related to PAD treatment and outcomes. The critical next step, therefore, is to create such tools and pilot their implementation as a foundation for broader integration of precision medicine and shared decision-making in clinical care.

Shared decision-making takes into account the latest evidence about all available treatment options and their outcomes, as well as patients' values and preferences with regards to treatment and potential outcomes that matter to them. Shared decision-making is extremely useful in treatment situations where there is clinical equipoise and where the choice of treatment should be greatly influenced by patients' preferences. Decision aids that facilitate this process of shared decision-making, have been consistently associated with better knowledge about the disease and treatments, less decisional conflict, and potential cost savings due to less invasive options being preferred by patients.

ELIGIBILITY:
Inclusion Criteria:

* All race and ethnicity categories, English speaking, men and women
* Age ≥18 years
* New onset complaints of PAD symptoms or exacerbation of previous PAD symptoms
* The diagnostic enrollment criterion includes a positive result for one of the following
* Doppler resting ankle-brachial index (ABI)≤0.90 or a significant drop in post exercise ankle pressure of ≥20 mmHg.
* Duplex
* CTA
* MRA
* TCOM
* Angiogram

Exclusion Criteria:

* Non-compressible ankle-brachial index (ABI ≥ 1.30)
* A lower limb revascularization procedure in the ipsilateral leg (same leg) where the patient is currently having symptoms in the past year (atherectomy, endarterectomy, bypass surgery, angioplasty)
* Peripheral intervention that occurs before the baseline interview
* Current episode of critical limb ischemia (ischemic rest pain, ulceration or gangrene) (Fontaine III, IV or Rutherford IV-VI)
* Patients with dementia
* Patients who are prisoners
* Patients who are unable to provide informed consent
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-06-24 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict | 6 months
  The primary outcome of this study will be decisional conflict as measured by the Decisional Conflict Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kim G Smolderen, PhD, Principal Investigator — University of Missouri Kansas City; Saint Luke's Hospital
Locations (1):
- Saint Luke's Hospital of Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] de Graaff JC, Ubbink DT, Kools EI, Chamuleau SA, Jacobs MJ. The impact of peripheral and coronary artery disease on health-related quality of life. Ann Vasc Surg. 2002 Jul;16(4):495-500. doi: 10.1007/s10016-001-0121-9. Epub 2002 Jun 27. PMID 12085126
- [Background] Rooke TW, Hirsch AT, Misra S, Sidawy AN, Beckman JA, Findeiss LK, Golzarian J, Gornik HL, Halperin JL, Jaff MR, Moneta GL, Olin JW, Stanley JC, White CJ, White JV, Zierler RE; Society for Cardiovascular Angiography and Interventions; Society of Interventional Radiology; Society for Vascular Medicine; Society for Vascular Surgery. 2011 ACCF/AHA Focused Update of the Guideline for the Management of Patients With Peripheral Artery Disease (updating the 2005 guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2011 Nov 1;58(19):2020-45. doi: 10.1016/j.jacc.2011.08.023. Epub 2011 Oct 6. No abstract available. PMID 21963765
- [Derived] Smolderen KG, Pacheco C, Provance J, Stone N, Fuss C, Decker C, Bunte M, Jelani QU, Safley DM, Secemsky E, Sepucha KR, Spatz ES, Mena-Hurtado C, Spertus JA. Treatment decisions for patients with peripheral artery disease and symptoms of claudication: Development process and alpha testing of the SHOW-ME PAD decision aid. Vasc Med. 2021 Jun;26(3):273-280. doi: 10.1177/1358863X20988780. Epub 2021 Feb 25. PMID 33627058